CLINICAL TRIAL: NCT01489475
Title: Plasma Angiopoietin Levels in Children Undergoing Modified Ultrafiltration Following Cardiopulmonary Bypass
Brief Title: Plasma Angiopoietin Levels in Children Following Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1107008778
Record Dates: First submitted 2011-11-29; First posted 2011-12-09 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2013-10

CONDITIONS: Congenital Heart Defects
Keywords: children; congenital heart defects; cardiopulmonary bypass; modified ultrafiltration; angiopoietins; cytokines
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Modified ultrafiltration fluid
  2. Whole blood which will be spun down to plasma (cells to be discarded)
Oversight: Data Monitoring Committee: No

SUMMARY:
During cardiopulmonary bypass (CPB) after heart surgery, a child's blood is exposed to many foreign entities. These conditions trigger the body's inflammatory response which results in leaky capillaries, increased swelling and possibly organ dysfunction. Since the early 1990's, modified ultrafiltration (MUF) has been shown to decrease excess swelling, reduce bleeding, improve heart function, and decrease hospital length of stay. Angiopoietins are a family of proteins necessary for both normal and abnormal blood vessel formation. They also appear to play a role in capillary leak. Though MUF has been shown to improve clinical outcome following CPB, there continues to be conflicting reports whether this is a result of the filtration of inflammatory proteins or simply from excess fluid removal. Since angiopoietins appear to play a role in both inflammation and capillary leak, the investigators hypothesize that the benefit seen after MUF is also secondary to its ability to filter out these proteins, especially angiopoietin-2.

DETAILED DESCRIPTION:
During cardiopulmonary bypass (CPB) for corrective or palliative congenital heart surgery, a child's blood is subjected to hemodilution, hypothermia, nonpulsatile blood flow and exposure to foreign and non-endothelialized surfaces. These non-physiologic conditions trigger the host's innate systemic inflammatory response which results in capillary leak, increased total body water and can lead to end organ dysfunction. Since the early 1990's, modified ultrafiltration (MUF) has been shown to decrease excess tissue edema, reduce postoperative bleeding, improve cardiac contractility, maintain hemodynamic stability, and decrease hospital length of stay. Angiopoietins are a family of vascular growth factors necessary for both normal and abnormal blood vessel formation and appear to play a role in capillary leak. Though MUF has been shown to improve clinical outcome following CPB, there continues to be conflicting reports whether this is a result of the filtration of inflammatory cytokines or simply excess fluid removal. Since angiopoietins appear to play a role in both inflammation and capillary leak, the investigators aim to determine whether MUF's clinical benefit is also secondary to its ability to filter out these molecules, more specifically angiopoietin-2.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with congenital heart disease undergoing surgical intervention requiring cardiopulmonary bypass and modified ultrafiltration.

Exclusion Criteria:

* Any patients with congenital heart disease who will not require modified ultrafiltration.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with congenital heart disease, undergoing surgical intervention requiring cardiopulmonary bypass and modified ultrafiltration will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pro- and anti-inflammatory protein levels after modified ultrafiltration | baseline to completion of MUF, on average 2 hours
  Modified ultrafiltration (MUF) is the process after cardiopulmonary bypass during which a filtration unit is added and blood is filtered and returned back to the patient. The goal of this project is to evaluate the effect of MUF on concentrations of Angiopoietin-2 (Ang-2) and IL 8, two known pro-inflammatory markers involved in capillary leakage, as well as Ang-1 and IL 10, two anti-inflammatory mediators. Levels will be drawn prior to bypass, after MUF and at ICU admission.
Change from baseline in pro- and anti-inflammatory protein levels at ICU admission | baseline to ICU admission, on average 7 hours
  Modified ultrafiltration (MUF) is the process after cardiopulmonary bypass during which a filtration unit is added and blood is filtered and returned back to the patient. The goal of this project is to evaluate the effect of MUF on concentrations of Angiopoietin-2 (Ang-2) and IL 8, two known pro-inflammatory markers involved in capillary leakage, as well as Ang-1 and IL 10, two anti-inflammatory mediators. Levels will be drawn prior to bypass, after MUF and at ICU admission.

SECONDARY OUTCOMES:
Biomarker correlation with patient outcome | Duration of pediatric ICU admission, on average 7 days
  The biomarkers will be compared to the age of patient, type of surgery performed as well as to post procedure outcome measurements to see if specific protein levels correlate with patient outcomes.
Pro- and anti-inflammatory protein presence in ultrafiltration fluid | Upon MUF completion, on average 2 hours
  MUF fluid samples will be drawn following bypass. Ang-2, Ang-1, IL-8 and IL-10 levels will be measured to determine if present.

CONTACTS AND LOCATIONS:
Overall Officials: John S Giuliano, Jr, MD, Study Director — Yale University
Locations (1):
- Yale Children's Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Result] Lang SM, Syed MA, Dziura J, Rocco E, Kirshbom P, Bhandari V, Giuliano JS Jr. The effect of modified ultrafiltration on angiopoietins in pediatric cardiothoracic operations. Ann Thorac Surg. 2014 Nov;98(5):1699-704. doi: 10.1016/j.athoracsur.2014.06.053. Epub 2014 Sep 23. PMID 25258157